CLINICAL TRIAL: NCT00281372
Title: Association Between Sexual Dysfunction in Adults and Behavioral Dysfunctions in Achieving Proper Dental Care
Brief Title: Sexual Dysfunction and Dental Care
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Gila Bronner, sheba medical center
Other Study IDs: SHEBA-05-3982-ES-CTIL
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Dyspareunia; Hypoactive Sexual Desire Disorder; Erectile Dysfunction; Vaginismus
Keywords: sexual dysfunction; male; female; dental care; need of control
MeSH Terms: conditions — Dyspareunia; Sexual Dysfunctions, Psychological; Erectile Dysfunction; Vaginismus; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

SUMMARY:
Evaluation of sexual functioning of patients at the Sexual Medical Center, at Sheba Medical Center in Israel. Sexual functioning shall be compared with their dental behavior.

Hypothesis: a positive association will be found.

DETAILED DESCRIPTION:
Patients, male and female, age over 18, who apply to the Sexual Medical Center, at Sheba Medical Center will fill a battery of questionnaires regarding their sexual function and dental treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, over 18 years old, who come for sexual therapy/ counseling to the Sexual Medical Center, in Sheba Medical Center, Israel Partners or spouses of the above.

Exclusion Criteria:

* Patients who are already in the middle of treatment.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women, over 18 years old, who come for sexual therapy/ counseling to the Sexual Medical Center, in Sheba Medical Center, Israel Partners or spouses of the above.
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2006-02; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shif, Prof. MD, Principal Investigator — Dept. of Obstetricts and Gynecology, Sheba Medical Center, Israel